CLINICAL TRIAL: NCT03902210
Title: An Online Wellness Intervention for Bone Marrow Transplant Survivors
Brief Title: BMT Online Wellness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00009352
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Bone Marrow Transplant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Yoga (Experimental): The intervention will be 12-weeks in duration and will consist of a series of pre-approved online yoga classes (6 manufactured specifically for the cancer-afflicted patients instructed by Udaya yoga therapist, Jules Mitchell, MS). Patients will be asked to complete a minimum of 60 minutes per week of yoga practice with encouragement to do more if they can. All Udaya.com videos will include a proper warm-up, cool down, and closing mindfulness activity (i.e., message from yoga therapist, brief meditation, final relaxation). Qualified Udaya yoga instructors who collectively have over 200 years of training and experience will expertly instruct the online yoga classes. Participants will be instructed to view a safety handout (see yoga safety & modifications handout) before gaining access to the Udaya video library. Yoga therapist, Jules Mitchell and PIs Huberty and Palmer will pre-approve Udaya videos that are appropriate for this population.
  Interventions: Behavioral: Online Yoga
- Podcast (Placebo Comparator): The podcast control group will be asked to view 60 minutes per week of online podcast videos. The podcast videos will contain general cancer-related health education material. To match the online yoga group for time and attention, 60 minutes per week will be prescribed, however, participants will have the ability to view additional videos each week. Furthermore, participants will also track their podcast video viewing each week in a daily log (see podcast group weekly log) by recording each time they view a video, the video that they viewed, and how long they viewed the video.
  Interventions: Behavioral: Podcast

INTERVENTIONS:
Behavioral: Online Yoga — 60 minutes per week of online yoga through Udaya.com
  Arms: Online Yoga
Behavioral: Podcast — 60 minutes per week of podcasts
  Arms: Podcast

SUMMARY:
Specific aim #1: Assess feasibility (i.e., acceptability, practicality, demand, limited efficacy) of a home-based, online yoga intervention in patients following allogeneic stem cell transplant. Feasibility benchmarks will include: >70% satisfied with the intervention and >70% intending to continue participating in online yoga (i.e., acceptability); >70% of participants achieving an average of >42 min/week (70% of presceibed 60 min/week) of online yoga throughout the 12-week intervention (i.e., demand); >70% completing questionnaires across all four time points (i.e., practicality); at least small effect sizes of the intervention on physical function, fatigue, anxiety, sleep disturbance, social functioning, pain interference, depression, and quality of life as compared to a podcast control group (i.e., limited efficacy).

DETAILED DESCRIPTION:
Online Yoga Group: The intervention will be 12-weeks in duration and will consist of a series of pre-approved online yoga classes (6 manufactured specifically for the cancer-afflicted patients instructed by Udaya yoga therapist, Jules Mitchell, MS). Patients will be asked to complete a minimum of 60 minutes per week of yoga practice with encouragement to do more if they can. All Udaya.com videos will include a proper warm-up, cool down, and closing mindfulness activity (i.e., message from yoga therapist, brief meditation, final relaxation). Qualified Udaya yoga instructors who collectively have over 200 years of training and experience will expertly instruct the online yoga classes. Participants will be instructed to view a safety handout (see yoga safety & modifications handout) before gaining access to the Udaya video library. Yoga therapist, Jules Mitchell and PIs Huberty and Palmer will pre-approve Udaya videos that are appropriate for this population.

A 12-week yoga prescription utilized in previous online yoga studies in MPN patients will be used in the proposed study for BMT patients. The 12-week yoga prescription was designed to be safe and progressive for cancer patients. During the intervention, all classes will offer alternative poses, modifications, and use of props (i.e., yoga blocks and straps) in the instance poses are difficult for the participant (i.e., painful, irregular, uneven breath) and to ensure safety. In addition to specific instruction regarding form and safety, the yoga therapist will provide descriptions of each video that includes tips and modifications to poses (e.g., set the knee on your yoga mat if this feels more comfortable for you). Additionally, patients will also receive a yoga modifications handout outlining the contraindicated yoga poses with modifications (see yoga safety & modifications handout). This handout will include an exercise warning for patients that experience dizziness, lightheadedness or faintness, excessive shortness of breath, chest pain, and that they need to stop the activity and contact their health care professional immediately if these symptoms are experienced.

The participants will access their yoga prescription on the Udaya.com website using their provided username and password (see instruction document). Participants will be asked to participate in a total of at least 60 minutes of yoga and keep a log of their participation utilizing a daily log available through a REDCap link (see yoga group weekly log). For the entire study, participants will record in their log each time they participate in yoga, the class in which they participated, how long they practiced (start and stop time), their perceived exertion, and their perceived mindfulness. Research staff will provide a weekly reminder email at the beginning of each week encouraging participation in their weekly yoga (see weekly reminder emails). We will ask that participants follow the yoga prescription, but if participants feel they want to deviate from the prescription they have the option to participate in any videos assigned in previous weeks or in any of the additional videos included each week in the prescription.

Podcast Control Group: The podcast control group will be asked to view 60 minutes per week of online podcast videos. The podcast videos will contain general cancer-related health education material. To match the online yoga group for time and attention, 60 minutes per week will be prescribed, however, participants will have the ability to view additional videos each week. Furthermore, participants will also track their podcast video viewing each week in a daily log (see podcast group weekly log) by recording each time they view a video, the video that they viewed, and how long they viewed the video.

ELIGIBILITY:
Inclusion Criteria:

* 1) have received a bone marrow transplant 6 months ago
* 2) have a cancer diagnosis
* 3) no active infections
* 4) platelet count >50
* 5) answer "no" to all items on the Physical Activity Readiness Questionnaire (PAR-Q), or be willing to obtain a signed medical release from their physician in the case that a question is answered with a "yes"
* 6) have access to a desktop or laptop on a regular basis
* 7) have access to reliable internet
* 8) read and understand English
* 9) age 18 years or older
* 10) willing to be randomized to one of two groups

Exclusion Criteria:

* 1) Engagement in yoga in the past year
* 2) currently engage in ≥150 min/week of moderate-/vigorous-intensity physical activity on a weekly basis
* 3) have a history of syncope in last 2 months
* 4) have a history of recurrent falls (≥2 in 2 months)
* 5) Any planned change in pharmacologic intervention (i.e., new drug) during the study interval (i.e., 20 weeks)
* 6) have an Eastern Cooperative Oncology Group 3 (ECOG 3) questionnaire score greater than three
* 7) currently utilize Udaya.com
* 8) currently pregnant
* 9) currently reside outside of the United States of America

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Physical Function | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Physical Function Subscale. Raw scores can range from 4-20, with higher scores indicating better physical function.
Anxiety | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Anxiety Subscale. Raw scores range from 4-20, with higher scores indicating more anxiety.
Depression | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Depression Subscale. Raw scores range from 4-20, with higher scores indicating more depression.
Fatigue | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Fatigue Subscale. Raw scores range from 4-20, with higher scores indicating more fatigue.
Sleep Disturbance | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Sleep Disturbance Subscale. Raw scores range from 4-20, with higher scores indicating more sleep disturbance.
Ability to Participate in Social Roles and Activities | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Ability to Participate in Social Roles and Activities Subscale. Raw scores range from 4-20, with higher scores indicating a better ability to participate in social roles and activities.
Pain Interference | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Pain Interference Subscale. Raw scores range from 4-20, with higher scores indicating more interference of pain in daily life.
Pain Intensity | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS-29 Pain Intensity Subscale. This is a single-item question asking the participant to rate their average level of pain on a 0-10 scale, with a higher score indicating worse pain.
Physical Health | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS Global Health Physical Subscale. Raw scores range from 2-10, with higher scores indicating better physical health.
Chronic Graft vs. Host Disease Symptoms | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured with the Lee Symptom Score, which assesses various symptoms commonly associated with Graft vs. Host Disease. Raw scores range from 0-120, with higher scores indicating higher symptom burden.
Mental Health | Change from baseline to midpoint (week 6), post-intervention (week 12), and follow-up (week 20)
  This measure is captured through the PROMIS Global Health Mental Health Subscale. Raw scores range from 2-10, with higher scores indicating better mental health.

SECONDARY OUTCOMES:
Objective Physical Activity | Daily physical activity throughout the 12-week intervention (baseline through week 12)
  Objective physical activity will be collected with the Fitbit Flex 2 device. This device captures light, moderate, and vigorous-intensity activity via an accelerometer.
Subjective Physical Activity | Weekly physical activity throughout the 12-week intervention (baseline through week 12)
  Subjective physical activity will be assessed with the Modifiable Activity Questionnaire. This questionnaire asks participants to indicate the days and the durations in which they participated in 39 different activities. Weekly minutes of activity is calculated from the information provided.
Objective Yoga/Podcast Participation | Weekly throughout the 12-week intervention (baseline through week 12)
  Participation in yoga or podcasts is collected through the number of minutes spent viewing/watching/listening to the yoga videos and podcast sessions.
Subjective Yoga/Podcast Participation | Weekly throughout the 12-week intervention (baseline through week 12)
  Participation in yoga or podcasts is collected through self-report yoga or podcast logs.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, Ph, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No